CLINICAL TRIAL: NCT02742857
Title: Non-randomized, Open-labeled, Interventional, Single Group, Proof of Concept Study With Multimodality Approach in Cases of Brain Death Due to Traumatic Brain Injury Having Diffuse Axonal Injury
Brief Title: Non-randomized, Open-labeled, Interventional, Single Group, Proof of Concept Study With Multi-modality Approach in Cases of Brain Death Due to Traumatic Brain Injury Having Diffuse Axonal Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioquark Inc. (Industry)
Collaborators: Revita Life Sciences (Unknown); Anupam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BQ12016; AAH -01-2016 (Other: Anupam Hospital)
Record Dates: First submitted 2016-04-06; First posted 2016-04-19 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Brain Death
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Biological: BQ-A Peptide Extract; Biological: Mesenchymal Stem Cells; Device: Transcranial Laser Therapy; Device: Median Nerve Stimulator

INTERVENTIONS:
Biological: BQ-A Peptide Extract — BQ-A Peptide Extract
Biological: Mesenchymal Stem Cells — Mesenchymal Stem Cells
Device: Transcranial Laser Therapy — Transcranial Laser Therapy
Device: Median Nerve Stimulator — Median Nerve Stimulator

SUMMARY:
This is the proof of concept study with multi-modality approach (using intra-thecal bioactive peptides, stem cells, laser and transcranial IV laser and Median Nerve stimulation as adjuvants) in cases of brain death due to traumatic brain injury having diffuse axonal injury to document possibility of reversal of brain death (BD).

ELIGIBILITY:
Inclusion Criteria:

* Individuals declared Brain dead from a traumatic brain injury having diffuse axonal injury on MRI
* Not willing for organ donation
* Written informed consent from the legally acceptable representative of the patient

Exclusion Criteria:

* Metallic clips/ metal implants or intracranial implants in the brain.
* Pregnancy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Reversal of brain death as noted in clinical examination or EEG | 15 days

SECONDARY OUTCOMES:
Cerebrospinal fluid (CSF) analysis of color consistency, cell counts, and microbial evaluation | 15 days
  To signify any signs of aseptic or bacterial meningitis
MRI analysis to analyze any changes in meninges | 15 days
  To signify any signs of aseptic or bacterial meningitis
Pulse | 15 days
O2 saturation | 15 days
Blood Pressure | 15 days
Respiration changes | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Himanshu Bansal, MD, Principal Investigator — Revita Life Sciences
Locations (1):
- Anupam Hospital, Rudrapur, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: Yes